CLINICAL TRIAL: NCT06557018
Title: Efficacy and Safety of Liposomal Bupivacaine Using Periarticular Injection for in Total Knee Arthroplasty: a Prospective, Randomized, Controlled Study
Brief Title: Efficacy and Safety of Liposomal Bupivacaine Using Periarticular Injection in Total Knee Arthroplasty
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dezhou Hospital Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DZSRMYYZC2023133
Record Dates: First submitted 2024-06-13; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- liposomal bupivacaine (LB) group (Experimental): 20cc liposomal bupivacaine (1 vial; 266 mg) added to 30 cc normal saline to a total of 50 cc solution was injected into the periarticular tissues at the conclusion of the surgical procedure.
  Interventions: Drug: liposomal bupivacaine
- traditional peri-articular injection group (Active Comparator): From periarticular injection consisted of 400 mg ropivacaine, 5 mg morphine and 0.4 mg epinephrine in 50 cc solution.
  Interventions: Drug: traditional peri-articular injection

INTERVENTIONS:
Drug: liposomal bupivacaine — liposomal bupivacaine group
  Arms: liposomal bupivacaine (LB) group
Drug: traditional peri-articular injection — traditional peri-articular injection group
  Other Names: Cocktail injection
  Arms: traditional peri-articular injection group

SUMMARY:
The goal of this clinical trial is to learn if drug Bupivacaine liposomes works better than traditional peri-articular injection for Control of Pain in Total Knee Arthroplasty. It will also learn about the safety of drug Bupivacaine liposomes.

The main questions it aims to answer are:

Does Bupivacaine liposomes works better than traditional peri-articular injection for Control of Pain in Total Knee Arthroplasty.

Researchers will compare Bupivacaine liposomes to traditional peri-articular injection to see if drug Bupivacaine liposomes works better for Control of Pain in Total Knee Arthroplasty

Participants will:

Receive peri-articular injection in total Knee Arthroplasty. checkups and tests During hospitalization.

DETAILED DESCRIPTION:
Total knee replacement (TKA) has made significant progress in the treatment of chronic intractable joint pain, and now the fastest effective way to treat serious knee diseases is to perform artificial knee replacement (TKA). Pain is an important factor affecting patients' satisfaction with TKA surgery, and it is also a key factor affecting patients' postoperative rehabilitation and reducing surgical complications.

Effective analgesia program can not only improve the postoperative satisfaction of patients, reduce the use of analgesic drugs, reduce postoperative adverse reactions, but also shorten the length of hospitalization and reduce hospitalization costs. Local Infiltration Analgesia (LIA) is a simple and effective analgesia technique that involves the infiltration of drugs into the wound during surgery. The duration of the analgesic effect can be prolonged by precisely placing the catheter at the surgical site for further local anesthesia after surgery. The most commonly used drugs for intra-articular and extra-articular injections are morphine, steroids, clonidine, epinephrine, ketorolac, ropivacaine, and bupivacaine.

Bupivacaine liposomes, as a new formulation of long-acting sustained-release bupivacaine, are of great significance for multimodal analgesia after TKA. At present, there are no studies on the application of bupivacaine liposomes and knee replacement in China. The purpose of this study was to observe the analgesic effect and effect on function of bupivacaine liposome used in local infiltration analgesia after total knee replacement, and to explore its analgesic effectiveness and safety, so as to provide some reference for the selection of analgesia for total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years.
2. American Society of Anesthesiologists (ASA) classification of grade I-II, with a certain level of literacy, good comprehension of Chinese language and text, no obstacles in doctor-patient communication, good understanding of visual analog scoring of pain (VAS scoring), and the ability to actively cooperate with the relevant examinations
3. Proposed initial unilateral total knee arthroplasty (TKA) under general anesthesia without any previous history of knee surgery.
4. The patients will participate in the study voluntarily, sign an informed consent form, and cooperate with all the assessments.

Exclusion Criteria:

1. Patients with other pain management options prior to surgery
2. Patients with neuromuscular pathology in the operated limb with other comorbidities that may affect postoperative recovery
3. Patients with allergy, hypersensitivity, intolerance, or contraindication to any of the drugs on study
4. Patients with a history of coronary artery, vascular stent placement, deep vein thrombosis, pulmonary embolism, myocardial infarction, or ischemic stroke treated within the past 6 months
5. The existence of serious liver and kidney dysfunction, coagulation disorders, cardiac arrhythmia, infection and other contraindications to surgery；
6. patients with any neurological or psychiatric disorders that may affect postoperative pain or interfere with study evaluation；
7. Patients with a history of misuse, abuse, or dependence on opioid analgesics, other prescription drugs, illicit drugs, or alcohol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
The VAS scores | 6 hours, 12 hours, 24 hours, 36 hours, 48 hours, 60 hours and 72 hours
  The VAS scores at 6 hours, 12 hours, 24 hours, 36 hours, 48 hours, 60 hours and 72 hours in the resting state and exercise state of the two groups were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Peilai Liu, Study Chair — Dezhou Hospital Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University Dezhou Hospital (Dezhou People's Hospital), Dezhou, Shandong, China

IPD SHARING:
Plan to Share IPD: No